CLINICAL TRIAL: NCT07138651
Title: Yoğun Bakım Hastalarına Uygulanan Aspirasyon Bakım Paketinin Ventilatör İlişkili Pnömoni Gelişimini Önlemeye Etkisi: Yarı Deneysel Çalışma
Brief Title: Effect of the Aspiration Care Bundle on Preventing VAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Banu Terzi, Assoc. Prof. Banu Terzi, Akdeniz University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2025/415
Record Dates: First submitted 2025-08-08; First posted 2025-08-24 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: VAP - Ventilator Associated Pneumonia; Care; Bundle Care; Aspiration; Nursing Care
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Intervention Model Description: A quasi-experimental study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Conrol group (Other): Rutin aspiration application
  Interventions: Other: Aspiration care bundle

INTERVENTIONS:
Other: Aspiration care bundle — Evidence-based aspiration care protocol

SUMMARY:
Many pharmacological and non-pharmacological interventions are used to prevent ventilator-associated pneumonia (VAP). Nurses are directly responsible for implementing non-pharmacological interventions and therefore have an important role in preventing VAP. The most important non-pharmacological nursing interventions to prevent VAP are hand hygiene and oral care. In addition, the head of the bed should be elevated to 30°-45°, head pressure should be monitored, and subglottic aspiration should be performed. Various care packages have been developed to prevent VAP. It has been determined that these care packages reduce the incidence of VAP. The aim of this study was to investigate the effect of the aspiration care package applied in the intensive care unit on preventing the development of ventilator-associated pneumonia, and it was planned as a quasi-experimental study.

DETAILED DESCRIPTION:
Ventilator-associated pneumonia (VAP) is defined as pneumonia that develops 48 hours after intubation in patients who did not have pneumonia at the time of intubation and who were placed on mechanical ventilation. VAP is known to be one of the most common healthcare-associated infections in patients admitted to intensive care units. VAP is a common nosocomial infection in intensive care units, and its consequences include high mortality, prolonged intensive care unit stay, and increased healthcare costs. There are two types of VAP: "early-onset" and "late-onset." Early-onset VAP develops 48-96 hours after intubation and is caused by microorganisms that are sensitive to antibiotic treatment. The microorganisms responsible for early-onset VAP include Methicillin-Sensitive Staphylococcus Aureus (MSSA), Streptococcus Pneumoniae, Haemophilus Influenzae, and Moraxella Catarrhalis. Late-onset VAP develops 96 hours after intubation and is caused by multidrug-resistant microorganisms. Microorganisms seen in late-onset VAP include Pseudomonas aeruginosa, methicillin-resistant Staphylococcus aureus (MRSA), Klebsiella species, and Acinetobacter baumannii. Clinical findings observed in patients with VAP include fever (body temperature above 38 degrees Celsius), leukocytosis (white blood cell count above 10,000 mm3), purulent secretion or increased secretion, and new or progressive infiltration on chest X-ray. Many pharmacological and non-pharmacological interventions are used to prevent VAP. Nurses are directly responsible for implementing non-pharmacological interventions and therefore have an important role in preventing VAP. The most important non-pharmacological nursing interventions to prevent VAP are hand hygiene and oral care. In addition, the head of the bed should be elevated to 30°-45°, head pressure should be monitored, and subglottic aspiration should be performed. Various care packages have been developed to prevent VAP. It has been determined that these care packages reduce the incidence of VAP. The aim of this study was to investigate the effect of the aspiration care package applied in the intensive care unit on preventing the development of ventilator-associated pneumonia, and it was planned as a quasi-experimental study.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the pulmonary intensive care unit
* Aged 18 years or older
* Connected to mechanical ventilation via ETT/TT
* Glasgow Coma Scale score: 8 or higher
* Remaining in the intensive care unit for at least 24 hours
* Patients who have not previously been diagnosed with ventilator-associated pneumonia will be included in the study.

Exclusion Criteria:

* Transferred from the pulmonary intensive care unit to another clinic
* Diagnosed with ventilator-associated pneumonia within the first 24 hours
* Glasgow Coma Scale score fell below 8 during the study
* Deceased at the time of data collection
* Patients who developed any complications related to aspiration (atelectasis, hypoxemia, bradypnea, etc.) prior to the study will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Clinical Pulmonary Infection Score | Through study completion, an average of 35 days
  Clinical Pulmonary Infection Score (CPIS):
  The CPIS is a clinical scoring system developed to facilitate the diagnosis of ventilator-associated pneumonia (VAP). It combines clinical, radiological, physiological, and microbiological parameters to provide a structured assessment of pulmonary infection in critically ill patients.
  Parameters evaluated in CPIS:
  * Temperature (fever or hypothermia)
  * Leukocyte count (leukocytosis, leukopenia, or normal range)
  * Tracheal secretions (absence, non-purulent, or purulent)
  * Arterial oxygenation (PaO₂/FiO₂ ratio)
  * Chest radiograph findings (infiltrates: absent, diffuse, or localized)
  * Culture of tracheal aspirate (no growth, light, or heavy growth of pathogenic bacteria) A total score >6 is commonly considered suggestive of pneumonia.
VAP rate monitoring form | Through study completion, an average of 35 days

IPD SHARING:
Plan to Share IPD: No